CLINICAL TRIAL: NCT04463615
Title: Pilot Trial of Leflunomide in Patients With CD30+ Lymphoproliferative Disorders
Brief Title: Leflunomide for the Treatment of Relapsed or Refractory CD30+ Lymphoproliferative Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19606; NCI-2020-02973 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 19606 (Other: City of Hope Medical Center); P30CA033572 (NIH)
Record Dates: First submitted 2020-07-06; First posted 2020-07-09 (Actual); Results first posted 2023-12-05 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-11

CONDITIONS: Recurrent Lymphoproliferative Disorder; Refractory Lymphoproliferative Disorder
MeSH Terms: conditions — Lymphoproliferative Disorders | interventions — Leflunomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (leflunomide) (Experimental): Patients receive leflunomide PO QD on days 1-28. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Leflunomide

INTERVENTIONS:
Drug: Leflunomide — Given PO
  Other Names: Arava; SU101

SUMMARY:
This trial studies how well leflunomide works for the treatment of patients with CD30+ lymphoproliferative disorders that have come back (relapsed) or do not respond to treatment (refractory). Leflunomide may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate overall response rate of leflunomide treatment.

SECONDARY OBJECTIVES:

I. To assess complete response rate and duration of response of leflunomide treatment.

II. To assess toxicities of leflunomide treatment. III. To assess disease status by the CAILS (composite assessment of index lesion severity).

EXPLORATORY OBJECTIVE:

I. To generate a preliminary ribonucleic acid (RNA) signature associated with response of CD30+ lymphoproliferative disorders (LYPDs) cells to leflunomide.

OUTLINE:

Patients receive leflunomide orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 13 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant and/or legally authorized representative

  * Assent, when appropriate, will be obtained per institutional guidelines
* Patients must have a life expectancy of > 3 months
* Eastern Cooperative Oncology Group (ECOG) =< 2
* Patients must have a diagnosis of cutaneous CD30+ LYPD
* Patients must be relapsed or are refractory to at least 1 prior line of therapy
* At least 2 weeks from prior therapy to time of start of treatment. Prior therapy includes steroids (except prednisone or equivalent - up to 10 mg/day is allowed)
* Absolute neutrophil count (ANC) >= 1000/mm^3 (within 21 days prior to day 1 of protocol therapy). NOTE: Growth factor is not permitted within 14 days of ANC assessment unless cytopenia is secondary to disease involvement
* Platelets >= 50,000/mm^3 (within 21 days prior to day 1 of protocol therapy). NOTE: Platelet transfusions are not permitted within 14 days of platelet assessment unless cytopenia is secondary to disease involvement
* Total bilirubin =< 1.5 X upper limit of normal (ULN) (unless has Gilbert's disease) (within 21 days prior to day 1 of protocol therapy)
* Aspartate aminotransferase (AST) =< 2.0 x ULN (within 21 days prior to Day 1 of protocol therapy)
* Alanine aminotransferase (ALT) =< 2.0 x ULN (within 21 days prior to day 1 of protocol therapy)
* Creatinine clearance of >= 30 mL/min per 24 hour urine test or the Cockcroft-Gault formula (within 21 days prior to day 1 of protocol therapy)
* Seronegative for human immunodeficiency virus (HIV) antigen (Ag)/antibody (Ab) combo, hepatitis C virus (HCV), active hepatitis B virus (HBV) (surface antigen negative) (within 21 days prior to day 1 of protocol therapy)

  * If positive, hepatitis C RNA quantitation must be performed
* Meets other institutional and federal requirements for infectious disease titer requirements. Note infectious disease testing to be performed within 28 days prior to day 1 of protocol therapy
* Negative for tuberculosis antigen (e.g. T-Spot test)
* Women of childbearing potential (WOCBP): negative urine or serum pregnancy test (within 21 days prior to day 1 of protocol therapy). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Agreement by females and males of childbearing potential* to use an effective method of birth control (hormonal or barrier method of birth control or abstinence) or abstain from heterosexual activity for the course of the study through at least three months after the last dose of protocol therapy. The effects of study treatment on a developing fetus have the potential for teratogenic or abortifacient effects. Should a woman become pregnant or suspect that she is pregnant while participating on the trial, she should inform her treating physician immediately

  * Childbearing potential defined as not being surgically sterilized (men and women) or have not been free from menses for > 2 years (women only)

Exclusion Criteria:

* Current or planned use of other investigational agents, or concurrent biological, chemotherapy, or radiation therapy during the study treatment period
* Current or planned growth factor or transfusion support. If growth factor or transfusion support is provided between screening and start of treatment, the participant will no longer be eligible
* Prior allogeneic transplant
* Acute active infection requiring systemic therapy within 2 weeks prior to enrollment
* Known history of hepatitis B or hepatitis C infection
* Known HIV infection
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to leflunomide or cholestyramine
* Non-hematologic malignancy within the past 3 years aside from the following exceptions:

  * Adequately treated basal cell or squamous cell skin cancer
  * Carcinoma in situ of the cervix
  * Prostate cancer < Gleason grade 6 with a stable prostate specific antigen (PSA)
  * Successfully treated in situ carcinoma of the breast
* Clinically significant medical disease or condition that, in the investigator's opinion, may interfere with protocol adherence or the patient's ability to give informed consent
* Pregnant women and women who are lactating. Leflunomide has potential for teratogenic or abortifacient effects. Because there is a potential risk for adverse events in nursing infants secondary to treatment of the mother with these agents, breastfeeding should be discontinued if the mother is enrolled on this study
* Any other condition that would, in the investigator's judgment, contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures, e.g., infection/inflammation, intestinal obstruction, unable to swallow medication, social/ psychological issues, etc
* Prospective participants who, in the opinion of the investigator, may not be able to comply with all study procedures (including compliance issues related to feasibility/logistics)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christiane Querfeld, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Leflunomide)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Leflunomide)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: Defined as the proportion of patients with a documented response (complete response [CR] or partial [PR]) any time during study treatment. Response will be categorized by modified severity weighted assessment tool (mSWAT). Will be calculated along with the Clopper Pearson binomial 95% exact confidence intervals. The treatment response was assessed after each 28-day cycle treatment.
Time Frame: Up to 42 days from the start time of the initial study treatment. Patient received one 28-day cycle treatment and then was off treatment on Day 14 of the second cycle due to disease progression.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Leflunomide)
Number analyzed (Participants) | 1
percentage of participants | 0

2. Secondary Outcome: Complete Response Rate
Description: Defined as the proportion of patients with a documented CR any time during study treatment. Response will be assessed by mSWAT. Will be calculated along with the Clopper Pearson binomial 95% exact confidence intervals. The treatment response was assessed after each 28-day cycle treatment.
Time Frame: Up to 42 days from the start time of the initial study treatment. Patient received one 28-day cycle treatment and was off treatment on Day 14 of the second cycle due to disease progression.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment (Leflunomide)
Number analyzed (Participants) | 1
percentage of participants | 0

ADVERSE EVENTS:
Time Frame: Up to 42 days from the start time of the initial study treatment. Patient received one 28-day cycle treatment and then was off treatment on Day 14 of the second cycle due to disease progression. The adverse effects were monitored and assessed at each cycle treatment. All-cause mortality monitored/assessed up to 84 days from the start time of the initial study treatment.
Arm/Group | Treatment (Leflunomide)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Leflunomide) (N=1)
Nausea (Gastrointestinal disorders) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT04463615/Prot_SAP_000.pdf